CLINICAL TRIAL: NCT03398681
Title: Changes in Myocardial Iron Content Following Administration of Intravenous Iron (Myocardial-IRON)
Brief Title: Changes in Myocardial Iron After Iron Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Julio Nuñez, Principal investigator, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYOCARDIAL-IRON; 2016-004194-40 (EudraCT Number)
Record Dates: First submitted 2017-11-21; First posted 2018-01-12 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Iron-deficiency
Keywords: Heart failure; Iron deficiency; Cardiac magnetic resonance; Ferric carboxymaltose; Myocardial iron
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Intervention Model Description: After providing informed consent, patients will be randomly assigned, with a remote, web-based computer-generated block randomization procedure in an allocation 1:1 ratio, to either receive intravenous ferric carboxymaltose (FCM) or placebo. Intramyocardial iron will be evaluated at 3 time points: before administration of CMF/placebo, and at 7 and 30 days. At 30 days, patients assigned to placebo will receive intravenous CMF if iron deficiency persists.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Because ferric carboxymaltose is a dark-brown solution that is easily distinguishable from the saline placebo, study personnel responsible for the preparation and administration of the study drug will aware of the group assignments and therefore, not involved in any study assessments. To ensure that patients will be unaware of the study drug, materials used in drug administration will be covered with aluminum foil or other opaque material and the injection site shield from the patient view. Once treatment is allocated, the investigators team will ensure that patients are blinded to the treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous ferric carboxymaltose (Active Comparator): Ferric Carboxymaltose solution [Ferinject® (FCM), Vifor Pharma (Glattbrugg, Switzerland)] will be given as a perfusion of 20 mL (which is the amount of FCM that is equivalent to 1000 mg of iron) diluted in a sterile saline solution (0.9% weight/volume (w/v) NaCl) administered over at least 15 min.
  Interventions: Drug: Ferric carboymaltose; Diagnostic Test: Cardiac magnetic resonance
- Normal saline (Placebo Comparator): Normal saline (0.9% weight/volume (w/v) NaCl) administered as per the instructions for active therapy.
  Interventions: Drug: Placebo (Normal saline); Diagnostic Test: Cardiac magnetic resonance

INTERVENTIONS:
Drug: Ferric carboymaltose — Ferric Carboxymaltose solution [Ferinject® (FCM), Vifor Pharma (Glattbrugg, Switzerland)]
  Other Names: Ferinject, intravenous iron
  Arms: Intravenous ferric carboxymaltose
Drug: Placebo (Normal saline) — Normal saline (0.9% weight/volume (w/v) NaCl)
  Arms: Normal saline
Diagnostic Test: Cardiac magnetic resonance — Cardiac magnetic resonance including T2* and T1-mapping sequences

SUMMARY:
Recent studies have shown that treatment with intravenous iron in patients with iron deficiency (ID) and heart failure with reduced ejection fraction (HFrEF) improves symptomatology, functional capacity, quality of life, and decreases hospitalizations regardless of anemia. In addition, a decrease in myocardial iron content has been observed in patients with chronic HFrEF. This preliminary evidence has led to postulate that myocardial iron deficiency could play a direct role in the pathogenesis and progression of the disease.

The investigators hypothesize that the repletion of myocardial iron would explain part of the benefit of this treatment. Thus, the investigators postulate that cardiac magnetic resonance (CMR) (T2* and T1-mapping sequences) will be sensible enough to detect changes in myocardial iron content as a result of intravenous iron administration, and that such changes will correlate with simultaneous changes in parameters of heart failure severity.

In this double-blind 1:1 randomized study controlled by placebo the investigators aim to determine the changes in myocardial iron content after treatment with intravenous ferric carboxymaltose (FCM) by CMR at 7 and 30 days in patients with stable HFrEF and ID.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ambulatory chronic heart failure
* Older than 18 years
* Patients in NYHA class II-III on optimal background therapy (as determined by the investigator) for at least 4 weeks with no dose changes of HF drugs during the last 2 weeks (with the exception of diuretics)
* Elevated natriuretic peptides levels (NT-proBNP >400 pg/ml) at the screening visit
* Left ventricle ejection fraction <50% documented in the last 12 months
* Iron deficiency defined as: serum ferritin level <100 μg/L or ferritin level 100-299 μg/L when TSAT is less than 20%, and hemoglobin <15 g/dL (all at screening)
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Known sensitivity to any of the products to be administered per protocol.
* History of acquired iron overload.
* Severe valve disease, or being scheduled for cardiac surgery within the next 30 days.
* Acute myocardial infarction or acute coronary syndrome, transient ischemic attack, or stroke within the last 3 months prior to randomization.
* Coronary artery bypass graft, percutaneous intervention (e.g. cardiac, cerebrovascular, and aortic; diagnostic catheters are allowed), or major surgery, including thoracic and cardiac surgery, within the last 3 months prior to randomization.
* Ischemic heart disease scheduled for revascularization procedures within the next 30 days.
* HF scheduled for cardiac resynchronization therapy within the next 30 days.
* Patients with active bleeding in the last 30 days.
* Known active infection or active malignancy.
* Subject at an immediate need of transfusion or hemoglobin ≥15 g/dL.
* Anemia due to reasons other than iron deficiency
* Immunosuppressive therapy or renal dialysis
* History of erythropoietin, intravenous iron therapy, and blood transfusion in the previous 12 weeks.
* Oral iron therapy at doses >100 mg/day in previous 1 week prior to randomization.
* Subjects with an immediate need for transfusion.
* Pregnant or breastfeeding women.
* Subject of childbearing potential who is not willing to use adequate contraceptive precautions during the study and for up to 5 days after the last scheduled dose of study medication.
* Subject currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study, or subject is receiving other investigational agent(s).
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in myocardial iron content assessed by CMR T2* | 7 and 30 days
Changes in myocardial iron content assessed by CMR T1-mapping | 7 and 30 days

SECONDARY OUTCOMES:
Changes in left ventricular systolic function evaluated with cardiac magnetic resonance | 7 and 30 days
  Changes in left ventricular systolic function evaluated with cardiac magnetic resonance
6-minute walking test | 7 and 30 days
  Changes in functional capacity assessed by distance walked in 6 minutes (6-minute walking test)
New York Heart Association (NYHA) class. | 7 and 30 days
  Changes in functional capacity assessed by New York Heart Association (NYHA) class.
The Kansas City quality of life questionnaire (KCCQ) | 7 and 30 days
  Quality of life assessed by The Kansas City quality of life questionnaire (KCCQ). KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Antigen carbohydrate 125 (CA125) | 30 days
  Laboratory tests, biomarkers: antigen carbohydrate 125 (CA125)
Amino-terminal pro-brain natriuretic peptide (NT-proBNP) | 30 days
  Laboratory tests, biomarkers: amino-terminal pro-brain natriuretic peptide (NT-proBNP)
Galectin-3 | 30 days
  Laboratory tests, biomarkers: galectin-3
ST-2 | 30 days
  Laboratory tests, biomarkers: ST-2
High-sensitivity troponin (hsTnT) | 30 days
  Laboratory tests, biomarkers: high-sensitivity troponin (hsTnT)
Cystatin C | 30 days
  Laboratory tests, biomarkers: cystatin C
Neutrophil gelatinase-associated lipocalin (NGAL) | 30 days
  Laboratory tests, biomarkers: neutrophil gelatinase-associated lipocalin (NGAL)
Serum creatinine | 30 days
  Laboratory tests: serum creatinine
Urea | 30 days
  Laboratory tests: urea
Estimated glomerular filtration rate (eGFR) | 30 days
  Laboratory tests: estimated glomerular filtration rate (eGFR)
Hemoglobin | 30 days
  Laboratory tests: hemoglobin
Ferritin | 30 days
  Laboratory tests: ferritin
Transferrin saturation (TSAT) | 30 days
  Laboratory tests: transferrin saturation (TSAT)
soluble transferrin receptor (sTfR) | 30 days
  Laboratory tests: soluble transferrin receptor (sTfR)
Hepcidin | 30 days
  Laboratory tests: hepcidin.
Clinical events: all-cause hospitalizations | 30 days
  All-cause hospitalizations
Clinical events: cardiovascular hospitalizations. | 30 days
  Cardiovascular hospitalizations
Clinical events: heart failure hospitalizations. | 30 days
  Heart failure hospitalizations
Clinical events: time to first hospitalization for any reason. | 30 days
  Time to first hospitalization for any reason.
Clinical events: time to first hospitalization for any cardiovascular reason. | 30 days
  Time to first hospitalization for any cardiovascular reason.
Clinical events: time to first hospitalization due to worsening heart failure. | 30 days
  Time to first hospitalization due to worsening heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Nuñez, MD PhD, Principal Investigator — Fundación Investigación Hospital Clínico Universitario de Valencia. Instituto de Investigación Sanitaria INCLIVA.
Locations (6):
- Spain (6):
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital de Manises, Manises, Valencia
  - ERESA, Valencia
  - Fundación Investigación Hospital Clínico Universitario de Valencia. Instituto de Investigación Sanitaria INCLIVA., Valencia
  - Hospital General de Valencia, Valencia
  - Hospital la Fe, Valencia

REFERENCES:
- [Derived] Del Canto I, Santas E, Cardells I, Minana G, Palau P, Llacer P, Facila L, Lopez-Vilella R, Almenar L, Bodi V, Lopez-Lereu MP, Monmeneu JV, Sanchis J, Moratal D, Maceira AM, de la Espriella R, Chorro FJ, Bayes-Genis A, Nunez J; Myocardial-IRON Investigators dagger. Short-Term Changes in Left and Right Ventricular Cardiac Magnetic Resonance Feature Tracking Strain Following Ferric Carboxymaltose in Patients With Heart Failure: A Substudy of the Myocardial-IRON Trial. J Am Heart Assoc. 2022 Apr 5;11(7):e022214. doi: 10.1161/JAHA.121.022214. Epub 2022 Mar 18. PMID 35301854
- [Derived] Meucci MC, Reinders MEJ, Groeneweg KE, Bezstarosti S, Ajmone Marsan N, Bax JJ, De Fijter JW, Delgado V. Cardiovascular Effects of Autologous Bone Marrow-Derived Mesenchymal Stromal Cell Therapy With Early Tacrolimus Withdrawal in Renal Transplant Recipients: An Analysis of the Randomized TRITON Study. J Am Heart Assoc. 2021 Dec 21;10(24):e023300. doi: 10.1161/JAHA.121.023300. Epub 2021 Dec 16. PMID 34913362
- [Derived] Nunez J, Minana G, Cardells I, Palau P, Llacer P, Facila L, Almenar L, Lopez-Lereu MP, Monmeneu JV, Amiguet M, Gonzalez J, Serrano A, Montagud V, Lopez-Vilella R, Valero E, Garcia-Blas S, Bodi V, de la Espriella-Juan R, Lupon J, Navarro J, Gorriz JL, Sanchis J, Chorro FJ, Comin-Colet J, Bayes-Genis A; Myocardial-IRON Investigators* dagger. Noninvasive Imaging Estimation of Myocardial Iron Repletion Following Administration of Intravenous Iron: The Myocardial-IRON Trial. J Am Heart Assoc. 2020 Feb 18;9(4):e014254. doi: 10.1161/JAHA.119.014254. Epub 2020 Feb 13. PMID 32067585
- [Derived] Minana G, Cardells I, Palau P, Llacer P, Facila L, Almenar L, Lopez-Lereu MP, Monmeneu JV, Amiguet M, Gonzalez J, Serrano A, Montagud V, Lopez-Vilella R, Valero E, Garcia-Blas S, Bodi V, de la Espriella-Juan R, Sanchis J, Chorro FJ, Bayes-Genis A, Nunez J; Myocardial-IRON Investigators. Changes in myocardial iron content following administration of intravenous iron (Myocardial-IRON): Study design. Clin Cardiol. 2018 Jun;41(6):729-735. doi: 10.1002/clc.22956. Epub 2018 Jun 5. PMID 29607528